CLINICAL TRIAL: NCT02837146
Title: Ultrasound Scores as Imaging Biomarkers of Early Response to Subcutaneous Tocilizumab in Association With Methotrexate in Very Early Rheumatoid Arthritis (TOVERA)
Brief Title: Ultrasound as Imaging Biomarker of Early Response to Tocilizumab and Methotrexate in Very Early Rheumatoid Arthritis
Acronym: TOVERA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Stoenoiu (Other)
Responsible Party: Sponsor-Investigator, Maria Stoenoiu, MD, PhD, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1200_14; 2015-001246-28 (EudraCT Number)
Record Dates: First submitted 2016-07-07; First posted 2016-07-19 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tocilizumab (TCZ) + Methotrexate (MTX) (Experimental): Induction phase:
  From week 0 to week 24, all subjects will receive TCZ and MTX
  Maintenance phase:
  From week 24 to week 54, all subjects will receive MTX
  Interventions: Biological: Tocilizumab (TCZ); Drug: Methotrexate (MTX)

INTERVENTIONS:
Biological: Tocilizumab (TCZ) — Induction phase: TCZ subcutaneously (162 mg weekly) from baseline to week 24
  Other Names: Ro-Actemra
Drug: Methotrexate (MTX) — Induction and maintenance phase: Methotrexate 15-20 mg/week from baseline to week 54
  Other Names: Ledertrexate, Emthexate

SUMMARY:
This study is aimed at assessing the kinetics of the ultrasound (US) response in DMARD-naive very early rheumatoid arthritis (RA) patients treated with tocilizumab (TCZ) and methotrexate (MTX).

DETAILED DESCRIPTION:
For most rheumatic autoimmune diseases, treatment has two components: induction of remission and maintenance (to prevent relapse). After screening (week -3 to 0), patients enter into a 3 week run-in period during which no glucocorticoid (GC) treatment is allowed. At week 0, if persistent synovitis is confirmed patients will enter the induction phase. During the induction phase all patients will receive TCZ and MTX from week 0 to week 24. After week 24, all patients will receive MTX.

Ultrasound (US) is increasingly used in rheumatic diseases, in particular in rheumatoid arthritis (RA). The great resolution of superficial musculoskeletal structures obtained by using high frequency transducers and the high sensitivity of colour Doppler (CD) and power Doppler (PD) techniques allow to detect synovial vascularisation, synovial hypertrophy (SH) and joint effusion (JE).

This is a pilot US trial that allow us to explore the hypothesis that an early US response may be predictive of later clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA fulfilling the 2010 EULAR/ACR (European League Against Rheumatism/ American College of Rheumatology classification criteria)
* Disease duration no longer than 12 months from the time of first swollen joint and no longer than 12 months from the time of initial diagnosis
* Age : 18-75 years
* Disease activity defined by a disease activity score DAS28-CRP > 3.2 or all must be met: tender joint count (TJC) of ≥4 and swollen joint count (SJC) ≥4
* US SH or PD synovitis scores >1 for at least 2 joints (MCP:2-5 or PIP:2-5 or CMC:2-5 or wrist joints or MTP:2-5 or ankle joints) and US SH or PD synovitis scores ≥1 for at least 1 other joint (MCP:2-5 or PIP:2-5 or or CMC:2-5 or wrist joints)
* Naïve to DMARDs (methotrexate, leflunomide, sulphasalazine) and naïve to any biologics or biosimilars.

Exclusion Criteria:

* History of other concomitant autoimmune disease such as lupus or psoriatic arthritis
* Meeting diagnostic criteria for any other rheumatic disease than RA (e.g. gout, Lyme disease, seronegative spondyloarthropathy including reactive arthritis, psoriatic arthritis, arthropathy or inflammatory bowel disease)
* Any previous treatment with :

  1. Biologics: Etanercept, infliximab, certolizumab, golimumab, abatacept, adalimumab, anakinra, tocilizumab, tofacitinib, etc.
  2. Any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti- CD3, anti-CD19 and anti-CD20
  3. Intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
  4. Alkylating agents such as chlorambucil, or with total lymphoid irradiation
* Previous MCP arthroplasty or wrist arthrodesis. Participants who have undergone or are scheduled to undergo joint arthroplasties other than the MCP joints can be recruited in the study provided all other eligibility criteria are met.
* Current liver disease requiring medication
* Current symptoms of severe progressive or uncontrolled renal, hematologic, gastro-intestinal, pulmonary, cardiac, neurologic or cerebral disease whether or not related to rheumatoid arthritis, that would jeopardize inclusion in the protocol as judged by the clinician
* History of malignancy or lymphoproliferative disease, within the last 5 years, with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma in situ of cervix which that has been fully excised/cured with no evidence of recurrence
* Concomitant diagnosis or history of diverticulitis, peptic ulcer disease, diverticulosis requiring antibiotic treatment or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis or other symptomatic lower GI conditions that might predispose to perforations
* Evidence of active or latent bacterial, viral, fungal (except for fungal infections of nail beds), mycobacterial or other opportunistic infections at the time of potential enrolment
* Any major episode of infection requiring hospitalisation or treatment with IV antibiotics within 4 weeks or oral antibiotics within 2 weeks of screening'
* Herpes zoster or cytomegalovirus infection that resolved less than 2 months before the informed consent was signed
* Subjects at risk of tuberculosis (TB) are excluded if any of the following is present:
* A history of active TB within the last 3 years, even if treated Latent TB that was not successfully treated ≥ 4 weeks Current clinical radiographic, or laboratory evidence of active TB
* Subjects who received live vaccines within 4 weeks of the anticipated first dose of study medication. Live and live attenuated vaccines should not be given concurrently
* Subjects must agree not to take live attenuated vaccines (including seasonal nasal flu vaccine, varicella vaccine for shingles or chickenpox, MMR or MMRV, oral polio vaccine and vaccines for yellow fever, measles, mumps or rubella) thirty (30) days before the Screening Visit, throughout the duration of the trial and for sixty (60) days following the subject's last dose of study drug
* Subjects with positive test results for hepatitis B surface antigen or hepatitis C, or HIV detected with polymerase chain reaction or immunoblot assay
* Subjects with primary or secondary immunodeficiency
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Major surgery within 8 weeks
* Patients with lack of peripheral venous access
* Pregnancy or breast-feeding
* Females of childbearing potential can only participate if using reliable contraception
* Intra-articular steroid injection in the joints assessed by US less than four weeks before screening
* Anticipated non-compliance with the protocol

Laboratory exclusion criteria

* Platelet count <100 x 109/l (100,000/mm3)
* Haemoglobin <85 g/l (8.5 g/dl; 5.3 mmol/l) (<8.0)
* White Blood Cells <3.0 x 109/l (3000/mm3) or >14,000/μl
* Absolute Neutrophil Count <2.0 x 109/l (2000/mm3)
* Absolute Lymphocyte Count <0.5 x 109/l (500/mm3)
* Positive Hepatitis BsAg, or Hepatitis C antibody
* Serum creatinine >1.4 mg/dl (124 μmol/l) in female patients and >1.6 mg/dl (141 μmol/l) in male patients. Patients with serum creatinine values exceeding limits may be eligible if their GFR is >30
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN)
* Total Bilirubin > ULN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in global ultrasound scoring system (GLOSS) at MCP (2-5 joints of both hands) and wrist joints | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54
  MCP=metacarpophalangeal; GLOSS scoring according to OMERACT: Grade 0 or normal=normal joint (no synovial hypertrophy (SH), no Doppler signal); Grade1 or minimal=minimal synovitis (minimal SH, with ≤ grade 1 Doppler signal); Grade 2 or moderate=moderate synovitis (moderate SH, with ≤ grade 2 Doppler signal or minimal SH and grade 2 Doppler signal); Grade 3 or severe=severe synovitis (severe SH with ≤ grade 3 Doppler signal or minimal or moderate SH and grade 3 Doppler signal). Joints are scored 0 to 3, and the sum of individual joints scores represents the total GLOSS for a subject.
The earliest time point at which improvement in GLOSS at MCP (2-5 joints of both hands) and wrists can be detected | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54

SECONDARY OUTCOMES:
GLOSS measured at 8 and 12 weeks is predictive to later clinical response at 24 and at 48 weeks | weeks 12, 24, 48
Minimum set of joints to be monitored by US in order to adequately assess disease activity | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54
Change in GLOSS for the whole US joint set | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54
Change in power Doppler (PD) scores for the whole US joint set | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54
Change in gray-scale (GS) scores for the whole US joint set | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54
Change in joint effusion (JE) scores for the whole US joint set | Baseline to weeks 2, 4, 8, 12, 16, 24, 32, 40, 54
Total PD score measured at 8 and 12 weeks is predictive to later clinical response at 24 and at 48 weeks | weeks 8, 12 , 24, 48
No radiographic progression assessed by Sharp/vdHeijde score | baseline to week 54
No new radiographic joint erosion at hands, wrists, ankles, feet | baseline to week 54
No new radiographic joint chondrolysis at hands, wrists, ankles, feet | baseline to week 54
No new swollen joint assessed by clinical examination | baseline to week 54
No new swollen joint assessed by ultrasound examination | baseline to week 54
DAS28 during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
SDAI during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
CDAI during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Swollen joint count score during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Tender joint count score for disease activity during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Patient visual analog score for disease activity during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Physician visual analog score for disease activity during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Number of patients fulfilling ACR/EULAR (2011) remission criteria during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Health assessment questionnaire(HAQ) score during the induction and maintenance phase | baseline to week 2, 4, 8, 12, 16, 24, 48, 54
Number of participants with serious adverse events(SAEs), with treatment-related SAEs, with discontinuations due to SAEs, with adverse events (AEs) with treatment-related AEs, with discontinuations due to AEs, death as outcome. | Days 1 to 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria S Stoenoiu, MD, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Maria S Stoenoiu, Brussels, Belgium, Belgium

IPD SHARING:
Plan to Share IPD: No